CLINICAL TRIAL: NCT03662113
Title: Effect of Domperidone on Completion Rate of Vedio Capsule Endoscopy: a Prospective Randomized Controlled Study
Brief Title: Effect of Domperidone on Completion Rate of Vedio Capsule Endoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Principal Investigator, Ying HUANG, The director of gastroenterology of Children's Hospital of Fudan University, Children's Hospital of Fudan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: DomperidoneVCE
Record Dates: First submitted 2018-09-04; First posted 2018-09-07 (Actual); Last update posted 2018-12-17 (Actual); Status verified 2018-12

CONDITIONS: Capsule Endoscopy; Pediatric Disorder
Keywords: domperidone
MeSH Terms: interventions — Domperidone; Simethicone; Water

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Domperidone (Experimental): 5ml domperidone prior to VCE
  Interventions: Drug: Domperidone
- Control: water (Other): 5ml warm water prior to VCE
  Interventions: Dietary Supplement: water

INTERVENTIONS:
Drug: Domperidone — 5ml Domperidone prior to VCE
  Other Names: simethicone
  Arms: Experimental: Domperidone
Dietary Supplement: water — 5ml water prior to VCE
  Other Names: simethicone
  Arms: Control: water

SUMMARY:
Video capsule endoscopy (VCE) has become an established technique to investigate the presence of small bowel pathology. But the limited battery life of capsules can lead to incomplete small bowel visualization. There is a rationale to use prokinetic agents prior to VCE reduce the chances of an incomplete small bowel examination via decrease gastric transit time (GTT). Investigators are aimed to prospectively compare the completion rate of VCE in pediatric patients receiving prokinetic with those receiving no prokinetic.

DETAILED DESCRIPTION:
Eligible children were randomly divided into two groups: domperidone prior to VCE and water prior to VCE. The primary outcome measure was the completion rate. Secondary outcome measures included the GTT and SBTT.

ELIGIBILITY:
Inclusion Criteria:

* Indications of capsule endoscopy;
* Informed consent form obtained.

Exclusion Criteria:

* Contraindication of capsule endoscopy;
* Domperidone allergy;
* Unwilling to participate.

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2018-11-01 (Actual)

PRIMARY OUTCOMES:
Completion rate of capsule endoscopy | assessed through study completion, an average of 1 year
  CE was considered complete when the cecum was reached within recording time.

SECONDARY OUTCOMES:
Gastric transit time (GTT) | assessed through study completion, an average of 1 year
  The GTT was defined as the time, in minutes, from the first image of the stomach until the first image of the duodenum.
small bowel transit time (SBTT) | assessed through study completion, an average of 1 year
  The SBTT was defined as the passage time, in minutes, from the first image of the duodenum until the first image of the cecum.

CONTACTS AND LOCATIONS:
Overall Officials: Ying Huang, doctor, Study Director — Children's Hospital of Fudan University
Locations (1):
- Children's hospital of Fudan university, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mcfarlane M, Liu B, Nwokolo C. Domperidone prolongs oral to duodenal transit time in video capsule endoscopy. Eur J Clin Pharmacol. 2018 Apr;74(4):521-524. doi: 10.1007/s00228-017-2399-8. Epub 2017 Dec 8. PMID 29222714
- [Derived] Wu J, Ye Z, Xue A, Huang Y. Can domperidone decrease transit time of pediatric video capsule endoscopy? A randomized controlled trial. Transl Pediatr. 2021 Feb;10(2):344-349. doi: 10.21037/tp-20-273. PMID 33708520